CLINICAL TRIAL: NCT05843825
Title: Effect of Using Block-out Spacer During Picking up of Locator Attachments Used for Retaining 3 Implant Mandibular Complete Overdenture: Peri-implant and Alveolar Bone Height Changes
Brief Title: Effect of Block-out Spacer to Pick up Locator Attachments to Retain Overdenture: Peri-implant and Alveolar Bone Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Rahma elhussany mohammed, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M11071020
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Bone Loss
Keywords: Peri-implant; Alveolar bone
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned into two equal groups . (BOS-G) Block out spacer group : patients who would be delivered mandibular implant overdenture retained by three locator attachments using block out spacer during pick up .(WBOS-G) Without block out spacer group : patients who would be delivered mandibular implant overdenture retained by three locator attachments without using block out spacer during pick up
Who Masked: Participant, Outcomes Assessor
Masking Description: The selected patients were stratified according to age, gender, years of mandibular edentulism, number of old non-satisfactory dentures.
  Patients were assigned to one of two groups using balanced randomization procedure to ensure comparability between groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (BOS-G) Block out spacer group (Active Comparator): (BOS-G)(Control group) : Patients who would be delivered mandibular overdenture retained by three locator attachments picked up using block out spacer .
  Interventions: Procedure: Surgical placement of dental implants; Device: Overdenture supported by locator attachment system
- (WBOS-G) Without block out spacer group (Active Comparator): (WBOS-G) (Study group): Patients who would be delivered mandibular overdenture retained by three locator attachments picked up without using block out spacer .
  Interventions: Procedure: Surgical placement of dental implants; Device: Overdenture supported by locator attachment system

INTERVENTIONS:
Procedure: Surgical placement of dental implants — Three dental implants were placed (one anterior in midline area and two posterior at first molar area).
Device: Overdenture supported by locator attachment system — Implants were loaded after three months by using locator attachments.
  Control group:Iocator attachments picked up using block out spacer.
  Study group:Iocator attachments picked up without using block out spacer

SUMMARY:
This study was conducted to radiographically evaluate peri-implant and alveolar bone height changes of locator attachments used for three implant assisted mandibular complete overdenture using two different pick up protocols.

DETAILED DESCRIPTION:
This clinical trial was done to evaluate the effect of using block-out spacer during picking up of locator attachments used for retaining 3 implant mandibular complete overdenture regarding peri-implant and alveolar bone height changes.

Eighteen egyptian completely edentulous male patients were chosen from the Outpatient Clinic of the Prosthodontics Department, Faculty of Dentistry, Mansoura University, Egypt.

Patients received three implants one anterior in midline area and two posterior at first molar area .

Patients free from any systemic diseases relating to the bone resorption, not taking any drugs that interfere with bone quality .Patients with absolute contraindication for surgical implantation, general contraindication , relative contraindication ,local contraindication for surgical implantation , allergic reactions to titanium or to local anesthesia were excluded.

The main question it aims to answer is whether to use block-out spacer during picking up of locator attachments used for retaining 3 implant mandibular complete overdenture or not.

* Participants were given antibiotic prophylaxis (clavulanic acid with amoxicillin 1 gm twice/day) one hour prior to surgery and continued for 6-7 days postoperative .Also, 50 mg of non-steroid anti-inflammatory tablets and analgesic (Declophenac tab) were given twice daily for one week after surgery. In addition to, Antiseptic mouth wash (0.2% chlorohexidine) was started ten minutes before surgery and continued one week after surgery twice daily.
* Patients were asked for radiographic evaluation immediately (T0) and 6 (T6) then 12 months (T12) after picking up of locator attachments.

Researcher compared between Block out spacer group (BOS-G) and Without block out spacer group (WBOS-G)which were randomly assigned into two equal groups to see if using block out spacer during picking up of locator attachments used for retaining 3 implant mandibular complete overdenture is more beneficial regarding peri-implant and alveolar bone height changes or not.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene practiced by edentulous patients.
* Completely edentulous maxillary and mandibular arches (at least six months since last extraction) .
* Mandibular residual alveolar ridge mucosa was healthy, firmly attached, well keratinized, free from any ridge flabbiness and even compressible mucosa as detected by palpitation with the blunt end of the mirror .
* Mandibular residual alveolar ridge form was U-shaped with accepted bone width, height and density as assessed by cone beam computed tomography.
* Angle's class I maxillo-mandibular relationship.
* Sufficient restorative space vertically not less than (8.5mm) and horizontally not less than (9 mm) which were verified by tentative jaw relation record and mounting on the articulator .

Exclusion Criteria:

* Systemic diseases relating to the bone resorption(e.g. osteoporosis , uncontrolled diabetes, osteogenesis imperfecta…etc).
* Administrated drugs that interfere with bone quality (e.g. corticosteroids, thyroxin, levothyroxine... etc).
* Patients with absolute contraindication for surgical implantation (recent myocardial infarction, cerebrovascular accident, valvular prosthesis surgery, immunosuppression, bleeding issues….etc).
* General contraindication for surgical procedures such as patient with head and neck radiotherapy and hepatic patients.
* Patients with relative contraindication: history of para functional habits such as bruxism, clenching and bad habits such as smoking and alcoholism .
* Local contraindication for surgical implantation (close proximity to vital structure, pathological lesion, remaining root not indicated for removal , localized bone defects or poor bone quality (D4)).
* Allergic reactions to titanium or to local anesthesia

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Peri-implant bone height changes (bone loss) | one year.
  Evaluations of vertical and horizontal peri-implant bone loss in mm by digital periapical radiography.

SECONDARY OUTCOMES:
Residual alveolar bone height changes (bone loss) | one year.
  Evaluations of vertical residual alveolar bone loss in mm by panoramic radiography.

CONTACTS AND LOCATIONS:
Overall Officials: Rahma El Hussany, MD, Principal Investigator — Mansoura University Faculty of Dentistry Prosthodontics Department
Locations (1):
- Rahma El Hussany, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No